CLINICAL TRIAL: NCT04760951
Title: Randomized Placebo-controlled Double-blinded Study of the Effect of TOTUM-070 on Lipid Metabolism in Moderate Hypercholesterolemic Subjects
Brief Title: Effect of Totum-070 on Lipid Metabolism in Moderate Hypercholesterolemic Subjects
Acronym: HEART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valbiotis (Industry)
Collaborators: Biofortis Mérieux NutriSciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PEC20070; 2020-A02809-30 (Other: ID-RCB)
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Hypercholesterolemia; Cardiovascular Risk Factor; Dyslipidemias; Overweight and Obesity; Atherosclerosis
Keywords: Moderate Hypercholesterolemia; Dyslipidemia; Overweight; Obesity; Cardiovascular Risk Factor; Nutrition Healthcare; Plant Extracts; Metabolic diseases; Atherosclerosis; Hygiene and dietary recommendations
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias; Overweight; Obesity; Atherosclerosis; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: 2 blinded arms (Active and Placebo)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TOTUM-070 (Experimental): Experimental active diet supplement TOTUM-070 taken 2 times per day
  Interventions: Dietary Supplement: TOTUM-070
- Placebo (Placebo Comparator): Placebo comparator taken 2 times per day
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: TOTUM-070 — 5-g dose of TOTUM-070 diet supplement, a mix of 5 plant extracts. Eight capsules per day to consume orally in two intakes
  Other Names: Active product
  Arms: TOTUM-070
Dietary Supplement: Placebo — Placebo. Eight capsules per day to consume orally in two intakes
  Other Names: Comparator product
  Arms: Placebo

SUMMARY:
This clinical study aims to assess the efficacy of TOTUM-070, a mix of 5 plant extracts, on lipid metabolism in moderate hypercholesterolemic subjects. The hypothesis is that TOTUM-070, daily consumed, is superior to placebo for decrease of fasting blood LDL-cholesterol concentration (determined by ultracentrifugation method) after 24 weeks of consumption.

ELIGIBILITY:
Inclusion Criteria:

* I1. From 18 to 70 years (including ranges);
* I2. Body mass index (BMI) between 18.5 and 35 kg/m² (including ranges);
* I3. Moderate hypercholesterolemic subject without any clinical symptoms of hypercholesterolemia (xanthoma, recurrent chest and/or leg pain) and not requiring immediate pharmacological lipid-lowering treatment according to the current recommendations (ESC/EAS, 2019);
* I4. For women: Non-menopausal with the same reliable contraception since at least three months before the beginning of the study and agreeing to keep it during the entire duration of the study (hormonal contraception, intra uterine device or surgical intervention) or menopausal with or without hormone replacement therapy (estrogenic replacement therapy begun from less than 3 months excluded);
* I5. Weight stable within ± 5% in the last three months;
* I6. No significant change in food habits or in physical activity in the 3 months before the randomization and agreeing to follow hygiene and dietary (HD) recommendations given during the study;
* I7. Good general and mental health according to the opinion of the investigator: no clinically significant and relevant abnormalities of medical history or physical examination;
* I8. Able and willing to participate to the study by complying with the protocol procedures as evidenced by his dated and signed informed consent form;
* I9. Affiliated with a social security scheme;
* I10. Agreeing to be registered on the volunteers in biomedical research.

At V0 biological analysis, the subjects will be eligible to the study on the following criteria:

* I11. Fasting blood LDL cholesterol concentration (using Friedewald estimation method) between 1.3 and 1.9 g/L (included ranges with ± 2% tolerated around);
* I12. Fasting blood triglycerides concentration ≤ 2.2 g/L;
* I13. SCORE Cardiovascular Risk Chart < 5% (Low-risk regions of Europe).

Exclusion Criteria:

* E1. Suffering from a metabolic disorder such as diabetes, uncontrolled thyroidal trouble or other metabolic disorder needing a dose adjustment in drug intervention according to the professional recommendations;
* E2. Suffering from an uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg);
* E3. With a history of ischemic cardiovascular event;
* E4. Having undergone recent surgical procedure in the past 6 months or in the 6 months to come;
* E5. With a history of bariatric surgery;
* E6. Suffering from a severe chronic disease (e.g. cancer, HIV, renal failure, ongoing hepatic or biliary disorders, chronic inflammatory digestive disease, arthritis or other chronic respiratory trouble, etc.) or gastrointestinal disorders found to be inconsistent with the conduct of the study by the investigator (e.g. celiac disease);
* E7. For women: ongoing pregnancy (as evidenced by a positive test for β-HCG (Human Chorionic Gonadotropin), i.e. > 5 mUI/mL, realized at V0) or breastfeeding or finished since less than 6 months or intending to become pregnant within 7 months ahead;
* E8. Under cholesterol and/or lipid-lowering treatment (e.g. statins, fibrates, ezetimibe, bile acid sequestrants, niacin, etc.) or stopped less than 3 months before the inclusion visit V0;
* E9. Under medication which could affect blood lipid parameters (e.g. long-term corticosteroid systemic drug, systemic antibodies, androgen or enzyme inducer, etc) or stopped less than 3 months before the inclusion visit V0 (antihypertensive stable long-term treatment tolerated);
* E10. Regular intake of dietary supplements or "health foods", or products rich in plant stanol or sterol (like Pro-Activ® or Danacol® products), rich in long chain omega-3 fatty acids (especially soft gels containing fish oils), or in other substances intended to reduce cholesterol or glycemia or stopped less than 3 months before the inclusion visit V0;
* E11. Under treatment or dietary supplement which could significantly affect parameter(s) followed during the study according to the investigator or stopped in a too short period before the randomization (for example consumed in the month before the randomization);
* E12. With a known or suspected food allergy or intolerance or hypersensitivity to any of the study products' ingredient;
* E13. Consuming more than 3 standard drinks daily of alcoholic beverage for men or 2 standard drinks daily for women or not agreeing to keep his alcohol consumption habits unchanged throughout the study;
* E14. With extreme eating habits (e.g. skipping meals regularly) or with a current or planned in the next 7 months specific diet (e.g. hyper or hypocaloric, vegan, vegetarian) or stopped less than 3 months before the study;
* E15. With a personal history of anorexia nervosa, bulimia or significant eating disorders according to the investigator;
* E16. Smoking more than 10 cigarettes daily or not agreeing to keep his smoking habits unchanged throughout the study. The subject should be able not to smoke the morning and during the visits;
* E17. Having a lifestyle deemed incompatible with the study according to the investigator including high level of physical activity (defined as more than 10 hours of intense physical activity a week, walking excluded);
* E18. Who made a blood donation in the 3 months before the randomization or intending to make it within 7 months ahead;
* E19. Taking part in another clinical trial or being in the exclusion period of a previous clinical trial;
* E20. Having received, during the last 12 months, indemnities for clinical trial higher or equal to 4500 Euros;
* E21. Under legal protection (guardianship, wardship) or deprived from his rights following administrative or judicial decision;
* E22. Presenting a psychological or linguistic incapability to sign the informed consent;
* E23. Impossible to contact in case of emergency.

At V0 biological analysis, the subjects will be considered as non-eligible to the study on the following criteria:

* E24. Fasting glucose plasma concentration > 126 mg/dL;
* E25. Blood AST (ASpartate amino Transferase), ALT (ALanine amino Transferase) or GGT (Gamma Glutamyl Transpeptidase) > 3 x ULN (Upper Limit of Normal);
* E26. TSH (Thyroid Stimulating Hormone) outside the laboratory normal values;
* E27. Blood urea > 12.11 mmol/L and/or creatinine concentration > 125 μmol/L;
* E28. Blood hsCRP > 10 mg/L;
* E29. Complete blood count (CBC) with hemoglobin < 11 g/dL or leucocytes < 3000 /mm3 or leucocytes > 16000 /mm3 or clinically significant abnormality according to the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Fasting blood LDL cholesterol concentration at V3 with ultracentrifugation method | V3 (24 weeks of intervention)
  Fasting blood LDL concentration (in g/L) with ultracentrifugation method, TOTUM-070 vs placebo

SECONDARY OUTCOMES:
Evolution of the fasting blood LDL cholesterol concentration with ultracentrifugation method | V1 (baseline) and V2 (12 weeks of intervention)
  Fasting blood LDL cholesterol concentration (in g/L) with ultracentrifugation method, TOTUM-070 vs placebo
Evolution of the fasting blood concentration of triglycerides | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Triglycerides (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of total cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Total cholesterol (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of HDL cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  HDL cholesterol (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of non-HDL cholesterol | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  non-HDL cholesterol (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of LDL cholesterol (Friedewald method) | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  LDL cholesterol (in g/L, Friedewald method), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of free fatty acids | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Free fatty acids (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood glycemia | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Glycemia (in mg/dL), TOTUM-070 vs placebo
Evolution of the fasting blood hsCRP concentration | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  hsCRP (in mg/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of apolipoprotein-A1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Apolipoprotein-A1 (in g/L), TOTUM-070 vs placebo
Evolution of the fasting blood concentration of apolipoprotein-B | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Apolipoprotein-B (in g/L), TOTUM-070 vs placebo
Evolution of atherogenic index | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Atherogenic index, TOTUM-070 vs placebo
Evolution of atherogenic coefficient | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Atherogenic coefficient, TOTUM-070 vs placebo
Evolution of Cardiac risk ratio 1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Cardiac risk ratio 1, TOTUM-070 vs placebo
Evolution of Cardiac risk ratio 2 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Cardiac risk ratio 2, TOTUM-070 vs placebo
Evolution of Apo-B/Apo-A1 ratio | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Apo-B/Apo-A1 ratio, TOTUM-070 vs placebo
Evolution of the body weight | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Body weight (in kg), TOTUM-070 vs placebo
Evolution of the waist circumference | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Waist circumference (in cm), TOTUM-070 vs placebo
Evolution of the hip circumference | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Hip circumference (in cm), TOTUM-070 vs placebo
Evolution of the waist to hip ratio | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Waist to hip ratio, TOTUM-070 vs placebo
Delay of occurence of pharmacological treatment requirement for hypercholesterolemia from V1 | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Delay between V1 and the date at which the investigator will decide to withdraw the subject from the study because he needs a pharmacological treatment to treat his hypercholesterolemia, TOTUM-070 vs placebo
Evolution of the cardiovascular disease risk (SCORE value) | V1 (baseline), V2 (12 weeks of intervention) and V3 (24 weeks of intervention)
  Systematic Coronary Risk Estimation value from Heartscore calculator

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Metreau, MD, Principal Investigator — Biofortis Mérieux NutriSciences
Locations (4):
- France (3):
  - Institut Pasteur de Lille, Lille
  - Unité d'Investigation Clinique Biofortis Mérieux NutriSciences, Paris
  - Biofortis Mérieux NutriSciences, Saint-Herblain
- Biotesys, Esslingen am Neckar, Germany

IPD SHARING:
Plan to Share IPD: No